CLINICAL TRIAL: NCT02791308
Title: Double-Blind Randomized Vehicle Controlled Study Evaluating Safety and Bioequivalence of Generic Pimecrolimus Cream 1% and Elidel® Comparing Both Active Treatments to a Vehicle Control in Treatment of Mild to Moderate Atopic Dermatitis
Brief Title: Study of Equivalence of Generic Pimecrolimus Cream 1% and Elidel® 1% in Subjects With Mild to Moderate Atopic Dermatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYM 2014-03
Record Dates: First submitted 2016-06-01; First posted 2016-06-06 (Estimated); Results first posted 2020-04-24 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — pimecrolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Pimecrolimus Cream, 1% (Experimental): Pimecrolimus Cream, 1% (Actavis)
  Interventions: Drug: Pimecrolimus Cream, 1%
- Elidel Cream, 1% (Active Comparator): Reference listed drug: Elidel 1% cream (Valeant Pharmaceuticals North America LLC)
  Interventions: Drug: Pimecrolimus Cream 1% (Valeant)
- Vehicle Cream (Placebo Comparator): Cream vehicle of the test product (Actavis)
  Interventions: Drug: Vehicle cream

INTERVENTIONS:
Drug: Pimecrolimus Cream 1% (Valeant)
  Other Names: Elidel® (pimecrolimus) Cream, 1% (Valeant)
  Arms: Elidel Cream, 1%
Drug: Vehicle cream
  Other Names: Vehicle of test product (Actavis)
  Arms: Vehicle Cream
Drug: Pimecrolimus Cream, 1%
  Other Names: Pimecrolimus Cream, 1% (Actavis)
  Arms: Pimecrolimus Cream, 1%

SUMMARY:
The purpose of this study is to compare the safety and efficacy profiles of Watson Laboratories, Inc.'s Pimecrolimus Cream, 1% to those of Valeant Pharmaceuticals North America LLC's Elidel® (pimecrolimus) Cream, 1%, and to demonstrate the superior efficacy of the two active creams over that of the placebo (Vehicle of test product), in the treatment of mild to moderate atopic dermatitis.

DETAILED DESCRIPTION:
Pimecrolimus cream, 1% is a calcineurin inhibitor immunosuppressant. Pimecrolimus inhibits T cell activation by blocking the transcription of early cytokines. Pimecrolimus cream, 1% is indicated as second-line therapy for the short-term and non-continuous chronic treatment of mild-to-moderate atopic dermatitis in non-immunocompromised adults and children 2 years of age and older who have failed to respond adequately to other topical prescription treatments, or when those treatments are not advisable. This study is being conducted to evaluate the clinical bioequivalence of sponsor's formulation of Pimecrolimus Cream, 1%, the Test product, and Elidel Cream, 1%, the Reference product. A vehicle control arm is included to demonstrate that the Test and Reference products are active and to establish that the study is sufficiently sensitive to detect differences between products.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent/assent for the study.
* Non-immunocompromised male or female aged 12 years or older.
* A clinical diagnosis of mild to moderate atopic dermatitis that has failed to respond adequately to other topical prescription treatments for atopic dermatitis, or subjects for whom the use of those other treatments is deemed inadvisable.
* A diagnosis of atopic dermatitis for at least 3 months.
* A baseline Investigator's Global Assessment (IGA) of disease severity of mild or moderate (score of 2 or 3).
* An affected area of atopic dermatitis involvement of at least 5% of the body surface area (BSA) at Visit 2/Day 1 (Baseline), as defined by the criteria of Hanifin and Rajka (1980).
* Treatment with a bland emollient for at least 7 days prior to Visit 2/Day 1 (Baseline).
* Agree to adhere to protocol-specified requirements and concomitant therapy restrictions.
* Willing to avoid constant sun exposure and the use of tanning booths or other UV light sources during participation in the study.
* In general good health, non-immunocompromised, and free from any clinically significant disease, other than atopic dermatitis, that might interfere with the study evaluations.
* Willing and able to understand and comply with the requirements of the study, apply the study medication as instructed, return for the required study visits, comply with therapy prohibitions, and complete the study.
* Female subjects of childbearing potential (excluding women who are surgically sterilized [hysterectomy, bilateral tubal ligation, or bilateral ovariectomy] or have been postmenopausal for at least 1 year) must have a negative urine pregnancy test and must be willing to use a medically accepted method of contraception during the study. The following are considered acceptable methods of birth control for the purpose of this study: oral contraceptives, contraceptive patches, contraceptive implant, vaginal contraceptive, double barrier methods (e.g., condom and spermicide), contraceptive injection (Depo-Provera®), intrauterine device (IUD), hormonal IUD (Mirena®), Essure® permanent birth control, and abstinence with a documented second acceptable method of birth control if the subject becomes sexually active. Subjects entering the study who are on hormonal contraceptives must have been on the method for at least 90 days prior to the study and continue the method for the duration of the study. Subjects who had used hormonal contraception and stopped must have stopped no less than 90 days prior to Visit 1.

Exclusion Criteria:

* Females who were pregnant, breastfeeding, intending to become pregnant during the study, or who did not agree to use an acceptable form of birth control during the study.
* Active cutaneous bacterial or viral infection in any proposed treatment area at Visit 2/Baseline (e.g., clinically infected atopic dermatitis).
* Sunburn, extensive scarring, or pigmented lesion(s) in any treatment area at Visit 2/Baseline that would interfere with the study evaluations.
* History of confounding skin conditions, e.g., psoriasis, rosacea, erythroderma, or ichthyosis.
* History or presence of Netherton's Syndrome, immunological deficiencies or diseases, HIV, diabetes, malignancy, serious active or recurrent infection, clinically significant severe renal insufficiency, or severe hepatic disorders.
* Use of any treatment listed in Table 9.1 more recently than the indicated washout period prior to Visit 2/Baseline.
* Need or intent to continue to use any treatment listed in Table 9.1 during the current study.

Ages: 12 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 587 (Actual)
Dates: Start 2015-02; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beth Landis, Study Director — Senior Clinical Project Manager
Locations (53):
- United States (53):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - Clinical Research Center of Alabama, Birmingham, Alabama
  - Agave Clinical Research, LLC, Mesa, Arizona
  - Omni Dermatology/Physicians Research Group, LLC, Phoenix, Arizona
  - Northwest Arkansas Clinical Trials Center, PLLC, Rogers, Arkansas
  - MD Studies, Inc., Fountain Valley, California
  - Alliance Research Centers, Laguna Hills, California
  - Medical Center for Clinical Research, San Diego, California
  - Skin Surgery Medical Group, Inc., San Diego, California
  - Horizons Clinical Research Ctr., LLC, Denver, Colorado
  - Immunoe International Research Centers, Thornton, Colorado
  - Dermatology of Boca, Boca Raton, Florida
  - Olympian Clinical Research, Clearwater, Florida
  - International Dermatology Research, Inc., Miami, Florida
  - Radiant Research, Inc., Pinellas Park, Florida
  - International Clinical Research- US, LLC, Sanford, Florida
  - MOORE Clinical Research, Inc., Tampa, Florida
  - Olympian Clinical Research, Tampa, Florida
  - Kansas City Dermatology PA, Overland Park, Kansas
  - Kentucky Pediatric/Adult Research, Bardstown, Kentucky
  - Dermatology Specialists Research, Louisville, Kentucky
  - Callender Center for Clinical Research, LLC, Glenn Dale, Maryland
  - David Fivenson, MD, PLC, Ann Arbor, Michigan
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - MediSearch Clinical Trials, Saint Joseph, Missouri
  - Quality Clinical Research Inc., Omaha, Nebraska
  - Karl G. Heine, MD Dermatology, Henderson, Nevada
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - Pinkas E. Lebovits, MD, PC, New York, New York
  - Piedmont Plastic Surgery and Dermatology, Charlotte, North Carolina
  - Dermatology Consulting Services, High Point, North Carolina
  - PMG Research of Winston-Salem, LLC, Winston-Salem, North Carolina
  - Cyn3rgy Research, Gresham, Oregon
  - Baker Allergy, Asthma and Dermatology Research Center, LLC, Portland, Oregon
  - Asthma & Allergy Research Associates, Upland, Pennsylvania
  - Clinical Partners, LLC, Johnston, Rhode Island
  - Greenville Dermatology, Greenville, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - ClinSearch, LLC, Chattanooga, Tennessee
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - J&S Studies, Inc., College Station, Texas
  - Suzanne Bruce and Associates, P.A./The Center for Skin Research, Houston, Texas
  - Center for Clinical Studies, Houston, Texas
  - Suzanne Bruce and Associates, P.A., The Center for Skin Research, Katy, Texas
  - R/D Clinical Research, Inc., Lake Jackson, Texas
  - Pflugerville Dermatology Clinical Research Center, Inc., Pflugerville, Texas
  - ACRC Trials, Plano, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - Intermountain Clinical Research, Draper, Utah
  - The Education and Research Foundation, Inc., Lynchburg, Virginia
  - National Clinical Research-Richmond, Inc., Richmond, Virginia
  - Dermatology Associates, Seattle, Washington
  - Eastern Washington Dermatology, Walla Walla, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Pimecrolimus Cream, 1%: Pimecrolimus Cream, 1% (Actavis)
  Pimecrolimus Cream, 1%
- Elidel Cream, 1%: Reference listed drug: Elidel 1% cream (Valeant Pharmaceuticals North America LLC)
  Pimecrolimus Cream 1% (Valeant)
- Vehicle Cream: Cream vehicle of the test product (Actavis)
  Vehicle cream
Period: Overall Study
Arm/Group | Pimecrolimus Cream, 1% | Elidel Cream, 1% | Vehicle Cream
Started | 195 | 196 | 196
Completed | 185 | 187 | 179
Not Completed | 10 | 9 | 17

BASELINE CHARACTERISTICS:
Population: Subjects included from Modified Intent-to-Treat Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Pimecrolimus Cream, 1% | Elidel Cream, 1% | Vehicle Cream | Total
Number analyzed (Participants) | 192 | 191 | 194 | 577
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.7 (18.16) | 37.4 (19.20) | 38.4 (18.61) | 36.8 (18.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116 | 107 | 115 | 338
  Male | 76 | 84 | 79 | 239
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 35 | 38 | 35 | 108
  Not Hispanic or Latino | 154 | 153 | 159 | 466
  Unknown or Not Reported | 3 | 0 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 1 | 4
  Asian | 13 | 21 | 16 | 50
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 63 | 60 | 68 | 191
  White | 101 | 100 | 99 | 300
  More than one race | 2 | 2 | 1 | 5
  Unknown or Not Reported | 11 | 7 | 9 | 27

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Treatment Success at Visit 4/Day 15
Description: Percentage of subjects in each treatment group with treatment success, defined as a grade of clear or almost clear (a score of 0 or 1 on the IGA) within all treatment areas at the end of treatment on Visit 4/Day 15
Time Frame: 15 days
Population: Per-Protocol Population
Measure: Count of Participants; unit: Participants
Arm/Group | Pimecrolimus Cream, 1% | Elidel Cream, 1% | Vehicle Cream
Number analyzed (Participants) | 164 | 162 | 156
Participants
  Success | 62 | 71 | 47
  Failure | 102 | 91 | 109
Statistical Analysis 1: Comparison: Pimecrolimus Cream, 1% vs Elidel Cream, 1%; Percentage of Subjects with Treatment Success at Visit 4/Day 15; Test type: Equivalence — Proportion of Subjects with Treatment Success at Visit 4/Day 15; Other = 0.407, 90% CI 2-sided [-15.57 to 3.53]

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Pimecrolimus Cream, 1% | Elidel Cream, 1% | Vehicle Cream
All-Cause Mortality (participants affected / at risk) | 0/192 | 0/191 | 0/194
Serious Adverse Events (participants affected / at risk) | 0/192 | 0/191 | 0/194
Other Adverse Events (participants affected / at risk) | 20/192 | 8/191 | 20/194
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pimecrolimus Cream, 1% (N=192) | Elidel Cream, 1% (N=191) | Vehicle Cream (N=194)
Eye Irritation (Eye disorders) | 1 | 0 | 0
Eye Swelling (Eye disorders) | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1
Application site hypersensitivity (General disorders) | 0 | 0 | 1
Application site pain (General disorders) | 1 | 0 | 1
Application site perspiration (General disorders) | 1 | 0 | 0
Application site pruritus (General disorders) | 1 | 0 | 1
Application site swelling (General disorders) | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 2
Cellulitis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Herpes Simplex (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 2 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 3 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0
Heachache (Nervous system disorders) | 3 | 1 | 0
Hypertonic bladder (Renal and urinary disorders) | 0 | 0 | 1
Breast tenderness (Reproductive system and breast disorders) | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1 | 5
Pruritis generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the study may be published or presented by the Investigator(s) after the review by, and in consultation and agreement with the Sponsor, and such that confidential or proprietary information is not disclosed.